CLINICAL TRIAL: NCT06588231
Title: Effect of Individualized Exercise Based on CPET on Multiple Cardiovascular Risk Factors and Cardiopulmonary Function in Elderly Patients With Coronary Heart Disease
Brief Title: Effect of Individualized Exercise in Elderly Patients With Coronary Heart Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Chen Leilei, Director, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IECHD
Record Dates: First submitted 2024-08-28; First posted 2024-09-19 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease | interventions — Clopidogrel; Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (Active Comparator): The patients in the control group were treated with routine rehabilitation nursing, while those in the control group were treated with routine antiplatelet drugs and lipid-lowering drugs after operation. Professional salesmen, according to the specific physical conditions of the patients, formulate corresponding recipes to ensure that the patients have a light diet, low salt, low fat and high nutritional value, and prohibit tobacco and alcohol.
  Interventions: Drug: optimal medical therapy ：aspirin, clopidogrel, statins.
- the exercise group (Experimental): The exercise group was given individualized rehabilitation training intervention on the basis of the control group. After 2 weeks of adaptive exercise training, there were no adverse events and voluntarily continued the participants. Under the guidance of the specialist, the exercise group received moderate and high intensity interval training, 3 times a week, 30-40 minutes each time, including the beginning of 5 minutes of warm-up and the last 5 minutes of cooling-off period.
  Interventions: Behavioral: Individual rehabilitation exercise training; Drug: optimal medical therapy ：aspirin, clopidogrel, statins.

INTERVENTIONS:
Behavioral: Individual rehabilitation exercise training — Under the guidance of a specialist, medium-and high-intensity interval training was conducted for 16 weeks, 3 times a week, 30-40 minutes each time, including the beginning of 5 minutes of warm-up and the last 5 minutes of cooling-off period, during which the exercise included 4 intervals, with the 85-95% pre intensity of HR reserve for 15-18 minutes, and then with the 50-70% pre intensity of HR reserve for 12-14 minutes, exercise for 3 minutes, and so on for 4 times. Warm-up and cooling-off periods can be done through stretching exercises, flexibility exercises (that is, neck, shoulders, upper back, buttocks and ankles) and low and medium intensity (50-70% heart rate reserve)
  Arms: the exercise group
Drug: optimal medical therapy ：aspirin, clopidogrel, statins. — those in the control group were treated with routine antiplatelet drugs and lipid-lowering drugs after operation. Professional salesmen, according to the specific physical conditions of the patients, formulate corresponding recipes to ensure that the patients have a light diet, low salt, low fat and high nutritional value, and prohibit tobacco and alcohol.
  Other Names: optimal medical therapy

SUMMARY:
The benefits of cardiac rehabilitation have been supported by a large amount of evidence-based medicine. Cardiac rehabilitation can correct cardiovascular risk factors, reduce morbidity and mortality, and improve quality of life.

DETAILED DESCRIPTION:
Cardiac rehabilitation includes drug, exercise, nutrition, psychological and behavioral intervention, smoking and alcohol restriction five prescription comprehensive medical measures, so as to improve the symptoms and prognosis of patients. Cardiac rehabilitation can not only delay the progress of the disease and improve the prognosis, but also improve the physical and mental state of patients, which has been recommended by the European Cardiology Association, the American Heart Association and the American Heart Association as Class I in the treatment of cardiovascular disease. Through the comprehensive intervention of patients, their physical, psychological and social functions can be restored to the best state, which can prolong life and significantly improve the quality of life, which is the essence of modern cardiac rehabilitation. Exercise rehabilitation is the core content of cardiac rehabilitation, which refers to the use of appropriate body exercise to help patients promote physical and mental health through exercise prescription and exercise guidance on the basis of comprehensive evaluation. The realization of sports rehabilitation requires a reasonable exercise prescription, which refers to the method of prescribing patients' exercise content and amount of exercise in the form of prescription according to individual physical condition and combining with environment and preference as far as possible. The best exercise prescription should be able to comprehensively promote health-related physical fitness, that is, cardiopulmonary endurance, muscle strength and endurance, flexibility, body composition and neuromotor fitness, and should be formulated in accordance with the principles of FITTVP, including frequency (several times a week), intensity (exertion), time (duration or total time), mode (pattern or type), as well as total and progress.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease: coronary angiography confirmed patients with coronary heart disease.
* Age is 60-75 years old, and the clinical sinus rhythm is stable.
* Left ventricular ejection fraction was> 40%.
* Informed consent and voluntary participation.

Exclusion Criteria:

* Patients with severe organic cardiac and lung diseases.
* Patients with hemiplegia and other physical action disorders.
* A history of mental illness.
* Uncontrolled hypertension, and hemodynamic instability.
* Severe nephropathy and severe peripheral artery disease.
* Patients with bone and joint diseases who are not suitable for exercise.
* Uncontrolled endocrine system and other diseases.
* Antibiotics and anti-diarrheal medications have not been used for at least 3 months.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-12-17 (Actual); Study Completion 2025-08-17 (Estimated)

PRIMARY OUTCOMES:
Gut microbiome | one year
  Fecal DNA isolation was performed using the QIA amp Fast DNA Stool Mini Kit (Qiagen, cat. 51604). After DNA extraction, fecal DNA was used for library preparation, and whole-genome shotgun sequencing was performed on the Illumina NovaSeq-6000 plat- form. From the raw metagenomic sequencing data, low-quality reads were discarded by the sequencing facility and reads belonging to human contaminations were removed by mapping the data to the reference genomes using Bowtie2. After filtering, on average, 54.8 million paired reads per sample were obtained for subsequent analysis.
Plasma metabolites profiles | one year
  Microbial metabolites profiles were generated using MetaPhlAn4 (version 4.0.3).
6MWT | one year
  6-minute walk test
LDL | one year
  low density lipoprotein
VO2peak | one year
  peak oxygen uptake

SECONDARY OUTCOMES:
Plasma metabolites concentration | one year
  The untargeted metabolome analysis was performed using an LC-MS/MS system.

CONTACTS AND LOCATIONS:
Overall Officials: Leilei Chen, Study Director — the First Affiliated Hospital of Nanjing Medical University, Nanjing, China
Locations (1):
- the First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No